CLINICAL TRIAL: NCT06657898
Title: Increasing Incidence of Complicated Pneumonia in Children in South-East Europe: a Retrospective Multi-center Analysis of Incidence, Characteristics and Outcomes
Brief Title: Complicated Pneumonia (CP) in Children in South-East Europe
Acronym: CP
Status: Recruiting | Type: Observational
Sponsor: Aleksandar Sovtic (Other)
Responsible Party: Sponsor-Investigator, Aleksandar Sovtic, Ass.Prof., Mother and Child Health Institute of Serbia Dr Vukan Cupic
Organization: Mother and Child Health Institute of Serbia Dr Vukan Cupic (Other)
Other Study IDs: CP-SEE-2024
Record Dates: First submitted 2024-10-01; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Pneumonia, Necrotizing; Lung Abscess; Empyema, Pleural
Keywords: pneumonia in children; necrotizing pneumonia; empyema; lung abscess
MeSH Terms: conditions — Pneumonia, Necrotizing; Lung Abscess; Empyema, Pleural; Empyema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective observational study aims to evaluate clinical course of complicated community acquired pneumonia in children, particularly focusing on necrotizing pneumonia cases, as well as determination of etiological agents (viruses and bacteria) and its association to severity and outcomes of the disease. Furthermore, therapeutic approach, complications, short-term and long-term outcomes and the prevention of the disease are to be assessed. The study will encompass data from pediatric centers in the South-East Europe willing to participate in the study, encompassing ten-year period of time.

DETAILED DESCRIPTION:
Children aged from 1 month to 18 years of age diagnosed with complicated community acquired pneumonia (pneumonia with parapneumonic effusion, necrotizing pneumonia or lung abscess) who were admitted from January 1st 2014 to April 30th 2024 to participating centers will be considered eligible for this multi-centric retrospective study.

The medical charts of all selected patients will be reviewed by medical professionals at each center and data collected in a standardized electronic database specifically created for this study to ensure consistency. Data quality will be internally monitored by the lead investigator, with periodic data validation checks to identify and resolve inconsistencies. All patient information will be stored securely in accordance with local regulations.

For every enrolled patient the following variables will be obtained: age, gender, date of admission, onset of symptoms and antibiotic treatment prior to hospitalization, comorbidities, immunization status, vital parameters on admission (heart rate, respiratory rate and percutaneous blood oxygen saturation), laboratory tests results on admission (white blood cells count, C-reactive protein concentration, blood gases, serum albumin concentration, serum lactate dehydrogenase activity), biochemical and cytological characteristics of pleural effusion (if applicable), microbiological results (culture and polymerase chain reaction) with Streptococcus pneumoniae serotype and its antimicrobial susceptibility to antibiotics, imaging (chest X-ray, CT scan, lung ultrasound), flexible bronchoscopy findings (if applicable), treatment modalities encompassing length of antibiotic therapy, use of systemic steroids, thoracic drainage, application of intrapleural fibrinolytics and surgical treatment, respiratory support information, length of hospitalization and intensive care unit stay, complications, chest radiography at follow up (at 3, 6, 12 months after discharge is available) and information on fatal/nonfatal outcome.

Primary outcome The primary outcome of this study is to estimate incidence and provide information on clinical characteristics of complicated community acquired pneumonia, particularly necrotizing pneumonia, in children and also identify possible association between microbiological isolates, immunization status and severity of clinical course.

Secondary outcomes

* Comparison of pre- and post- pneumococcal conjugate vaccine period (in selected countries) regarding the number of cases, isolated Streptococcus pneumoniae and antimicrobial resistance
* Determining if high values of inflammatory markers in serum can be predictive factors for complicated clinical course
* Evaluation of the effectiveness of the early introduction of intrapleural fibrinolytic therapy to length of hospital stay and incidence of complications (including bronchopleural fistula).
* Use the systemic corticosteroids for empyema and associated necrotizing pneumonia and the risk for bronchopleural fistula
* Evaluation of frequent use of antibiotics and higher prevalence of multi-drug resistant Streptococcus pneumoniae.
* Determination of risk factors for surgical therapy

The primary outcome, incidence of complicated community acquired pneumonia, will be compared between vaccinated and non-vaccinated groups using chi-square tests for categorical variables and t-tests for continuous variables. Secondary outcomes, such as length of hospital stay and complications, will be analyzed using ANOVA and logistic regression, adjusting for potential confounders such as age and comorbidities. Subgroup analyses will assess differences in outcomes across age groups and different vaccination periods (pre- and post- 13 valent pneumococcal conjugate vaccine). Statistical significance will be defined as p<0.05. Statistical analyses will be performed using SPSS, version 26.

ELIGIBILITY:
Inclusion Criteria

* Children aged 1 month to 18 years of age
* Children diagnosed with complicated community acquired pneumonia (pneumonia with parapneumonic effusion, necrotizing pneumonia and lung abscess)
* Children who were hospitalized from January 1st 2014 to April 30th 2024 and required at least 24 hours of hospital stay

Exclusion Criteria

* Children with increased risk for severe lung infections (cystic fibrosis, primary ciliary dyskinesia, immunodeficiencies, congenital lung abnormalities, neurological conditions, chemotherapy)
* Children with hospital-acquired pneumonia

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged from 1 month to 18 years of age diagnosed with complicated community acquired pneumonia (pneumonia with parapneumonic effusion, necrotizing pneumonia or lung abscess) and who were admitted from January 1st 2014 to April 30th 2024 in participating centers will be considered eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of children hospitalized and diagnosed with complicated (particularly necrotizing) community-acquired pneumonia relative to the total number of children hospitalized for community-acquired pneumonia over the study period and for each year | January 1st 2014 to April 30th 2024
  The values will be expressed as percentage. Incidence rates will be calculated for each year and across different centers.

SECONDARY OUTCOMES:
Distribution of different types of complicated community acquired pneumonia | from hospital admission to discharge, lasting on average from one to three weeks.
  The value will be collected as categorical variable (different category for each type: pleural effusion, necrotizing pneumonia, lung abscess). It will be expressed as percentage of total number of participants. Statistical analysis will be conducted in order to determine which types are related to longer hospitalization, ICU admission, more severe clinical course, fatal outcome, incomplete radiological resolution on follow ups and complications.
Number of participants vaccinated against Streptococcus pneumoniae with pneumococcal conjugate vaccine and distribution of vaccines covering for different number of serotypes | from hospital admission to discharge, lasting on average from one to three weeks.
  The value will be collected as categorical variable (categories for vaccinated and non-vaccinated). It will be expressed as percentage of total number of participants. Statistical analysis will be conducted in order to determine if non-vaccinated participants had longer hospitalization, ICU admission, more severe clinical course, fatal outcome, incomplete radiological resolution on follow ups and complications.
Distribution of different Streptococcus pneumoniae vaccines covering for different number of serotypes | from hospital admission to discharge, lasting on average from one to three weeks.
  The value will be collected as categorical variable (category for vaccines covering for different number of serotypes). It will be expressed as percentage of total number of participants vaccinated. Statistical analysis will be conducted in order to determine relation of vaccines covering for different serotypes with different Streptococcus pneumoniae serotype distribution, hospitalization length, ICU admission, more severe clinical course, fatal outcome, incomplete radiological resolution on follow ups and complications.
Duration of symptoms before hospitalization | recorded at the time of hospital admission.
  The value will be expressed as continuous variable (number of days). The duration of symptoms before hospitalization will be analyzed using descriptive statistics, reported as a mean (± standard deviation) and median (with interquartile range). Regression analysis may be used to identify factors associated with longer symptom duration (e.g., age, vaccination status). Comparison between groups of participants with different types of complicated community-acquired pneumonia will be done.
Percutaneous oxygen saturation (SpO2) | recorded at the time of hospital admission.
  The value will be collected as continuous variable in percentages, as well as categorical (level below and above 95%).
  It will be summarized using descriptive statistics (mean ± standard deviation for continuous variables, and frequencies for categorical data) and used as one of indicators of the severity of the disease. Comparison between groups of participants with different types of complicated community-acquired pneumonia, as well as vaccinated and non-vaccinated participants against Streptococcus pneumoniae, and different causative agents will be done.
  Logistic regression may be used to assess whether lower SpO2 on admission is associated with more severe clinical outcomes, ICU admission, longer hospitalization length, or complications.
Heart rate | recorded at the time of hospital admission.
  The value will be recorded as continuous variable as beats per minute. It will be summarized using descriptive statistics (mean ± standard deviation or median and interquartile range) and used as one of indicators of the severity of the disease. Comparison between groups of participants with different types of complicated community-acquired pneumonia, different vaccinal status and different causative agents will be done.
  Logistic regression may be used to assess whether elevated heart rate is associated with more severe clinical outcomes, ICU admission, longer hospitalization length, or complications.
Respiratory rate | recorded at the time of hospital admission.
  The value will be recorded as continuous variable as breaths per minute. It will be summarized using descriptive statistics (mean ± standard deviation or median and interquartile range) and used as one of indicators of the severity of the disease. Comparison between groups of participants with different types of complicated community-acquired pneumonia, different vaccinal status and different causative agents will be done.
  Logistic regression may be used to assess whether elevated respiratory rate is associated with more severe clinical outcomes, hospitalization length, ICU admission or complications.
White blood cells count | recorded at the time of hospital admission.
  The value will be recorded as continuous variable (number of cells x10^9 per liter).
  It will be summarized using descriptive statistics (mean ± standard deviation or median with interquartile range) and used as one of indicators of the severity of the disease. Comparison between groups of participants with different types of complicated community-acquired pneumonia, different vaccinal status and different causative agents will be done.
  Logistic regression may be used to assess whether elevated white blood cells count is associated with more severe clinical outcomes, longer hospitalization, ICU admission, surgical treatment or complications.
C-reactive protein concentration | recorded at the time of hospital admission.
  The value will be recorded as continuous variable (concentration in mg/L). It will be summarized using descriptive statistics (mean ± standard deviation or median and interquartile range) and used as one of indicators of the severity of the disease. Comparison between groups of participants with different types of complicated community-acquired pneumonia, different vaccinal status and different causative agents will be done.
  Logistic regression may be used to assess whether elevated concentration of C-reactive protein is associated with more severe clinical outcomes, longer hospitalization, ICU admission, surgical treatment or complications.
Blood serum albumin concentration | recorded at the time of hospital admission.
  The value will be recorded as continuous variable (expressed in g/L). It will be summarized using descriptive statistics (mean ± standard deviation or median and interquartile range) and used as one of indicators of the severity of the disease. Comparison between groups of participants with different types of complicated community-acquired pneumonia, different vaccinal status and different causative agents will be done.
  Logistic regression may be used to assess whether lower concentration serum albumin is associated with more severe clinical outcomes, longer hospitalization, ICU admission, surgical treatment or complications.
Serum lactate dehydrogenase activity | recorded at the time of hospital admission.
  The value will be recorded as continuous variable (expressed in IU/L). It will be summarized using descriptive statistics (mean ± standard deviation or median and interquartile range) and used as one of indicators of the severity of the disease and indicator of lung necrosis. Comparison between groups of participants with different types of complicated community-acquired pneumonia, different vaccinal status and different causative agents will be done.
  Logistic regression may be used to assess whether elevated serum activity of lactate dehydrogenase is associated with more severe clinical outcomes, longer hospitalization, ICU admission, surgical treatment or complications.
Positivity of pleural fluid bacteriological culture and PCR (polymerase chain reaction) to bacteria (if done) | from hospital admission to discharge, lasting on average from one to three weeks.
  The data will be collected as categorical variables (each category for different causative agent) and measured in order to provide potential causative for complicated community-acquired pneumonia.
  It will be expressed as a percentage of all participants tested and used for the comparison between groups of participants with different types of complicated community-acquired pneumonia. Frequency distribution of Streptococcus pneumoniae isolate will be compared between participants vaccinated and non-vaccinated against Streptococcus pneumoniae, and also between participants in periods of time regarding introduction of pneumococcal conjugate vaccine.
  It is also going to be evaluated if certain bacterial causatives are associated with more severe clinical outcomes, longer hospitalization, ICU admission, surgical treatment, fatal outcome or complications.
Positivity of blood bacteriological culture and PCR (polymerase chain reaction) to bacteria (if done) | from hospital admission to discharge, lasting on average from one to three weeks.
  The data will be collected as categorical variables (each category for different causative agent) and measured in order to provide potential causative for complicated community-acquired pneumonia.
  It will be expressed as a percentage of all participants tested and used for the comparison between groups of participants with different types of complicated community-acquired pneumonia. Frequency distribution of Streptococcus pneumoniae isolate will be compared between participants vaccinated and non-vaccinated against Streptococcus pneumoniae, and also between participants in periods of time regarding introduction of pneumococcal conjugate vaccine.
  It is also going to be evaluated if certain bacterial causatives are associated with more severe clinical outcomes, longer hospitalization, ICU admission, surgical treatment, fatal outcome or complications.
Positivity of bronchoalveolar lavage fluid bacteriological culture and PCR (polymerase chain reaction) to bacteria (if done) | from hospital admission to discharge, lasting on average from one to three weeks.
  The data will be collected as categorical variables (each category for different causative agent) and measured in order to provide potential causative for complicated community-acquired pneumonia.
  It will be expressed as a percentage of all participants tested and used for the comparison between groups of participants with different types of complicated community-acquired pneumonia. Frequency distribution of Streptococcus pneumoniae isolate will be compared between participants vaccinated and non-vaccinated against Streptococcus pneumoniae, and also between participants in periods of time regarding introduction of pneumococcal conjugate vaccine.
  It is also going to be evaluated if certain bacterial causatives are associated with more severe clinical outcomes, longer hospitalization, ICU admission, surgical treatment, fatal outcome or complications.
Positivity to viral causative agents on PCR (polymerase chain reaction) (if done) | from hospital admission to discharge, lasting on average from one to three weeks.
  The data will be collected as categorical variables (each category for different causative agent) and measured in order to provide potential causative for complicated community-acquired pneumonia.
  It will be expressed as a percentage of all participants tested and used for the comparison between groups of participants with different types of complicated community-acquired pneumonia.
  It is also going to be evaluated if certain bacterial causatives are associated with more severe clinical outcomes, longer hospitalization, ICU admission, surgical treatment, fatal outcome or complications.
Identification of specific Streptococcus pneumoniae serotype if isolated (if serotyping done) | from hospital admission to discharge, lasting on average from one to three weeks.
  The data will be recorded as categorical variables (each category for different serotype) and is collected to provide insight into Streptococcus pneumoniae serotype distribution.
  It will be expressed as percentage and used for the comparison between participants vaccinated and non-vaccinated against Streptococcus pneumoniae, as well as between participants who were immunized with pneumococcal conjugate vaccine covering for different number of serotypes. Also, the serotype distribution will be compared between participants in periods of time regarding introduction of pneumococcal conjugate vaccine. Comparison between groups of participants with different types of complicated community acquired pneumonia will be done, as well.
  Its relation to complications, surgical treatment, fatal outcome and incomplete radiological resolution on follow-ups will be analyzed.
Resistance of Streptococcus pneumoniae to penicillin and ceftriaxone, and resistance of Staphylococcus aureus to methicillin | from hospital admission to discharge, lasting on average from one to three weeks.
  The data will be recorded as categorical variables (two categories for each, resistant and sensitive).
  It will be expressed as percentage of all participants that had positive cultures to applicable bacteria and compared between groups of participants with and without use of antibiotics just prior to hospitalization.
Duration of antibiotic therapy (peroral and intravenous) | from hospital admission to discharge, lasting on average from one to three weeks, and at first follow-ups.
  The data will be recorded as continuous variables (number of days). It will be summarized using descriptive statistics (mean ± standard deviation or median and interquartile range). The data will be compared between groups of participants with different types of complicated community-acquired pneumonia, different vaccinal status and different causatives. Analysis will also be conducted in order to determine potential association between length of antibiotic therapy and incomplete resolution on follow ups.
Use of systemic corticosteroids | from hospital admission to discharge, lasting on average from one to three weeks.
  The data will be recorded as categorical variables (corticosteroids administered and not administered).
  It will be expressed as percentage of all participants. The data will be compared between groups of participants with different types of complicated community-acquired pneumonia, different vaccinal status and different causatives. Analysis will be conducted in order to determine potential association between steroid therapy length and occurrence of complications, especially bronchopleural fistula. Also, its relation to hospitalization length and potential association with surgical treatment, fatal outcome and incomplete radiological resolution on follow-ups will be analyzed.
Level of respiratory support | from hospital admission to discharge, lasting on average from one to three weeks.
  The data will be recorded as categorical variables (each category for different type of respiratory support being low flow oxygen therapy, high flow oxygen therapy, non-invasive mechanical ventilation and invasive mechanical ventilation) and is used as one of indicators of severity of the disease.
  It will be expressed as percentage. The data will be compared between groups of participants with different types of complicated community-acquired pneumonia, different vaccinal status and also different causative agents. Also, analysis will be conducted in order to determine its potential association with complications, surgical treatment, fatal outcome and incomplete radiological resolution on follow-ups.
Number of participants requiring pleural drainage | from hospital admission to discharge, lasting on average from one to three weeks.
  The data will be recorded as categorical variables (two categories, with and without pleural drainage), and is used as one of indicators of severity of the disease.
  It will be expressed as percentage of all participants. The data will be compared between groups of participants with different types of complicated community-acquired pneumonia, different vaccinal status and also different causative agents.
  Its relation to complications, surgical treatment, fatal outcome and incomplete radiological resolution on follow-ups will be analyzed.
Duration of pleural drainage | from hospital admission to discharge, lasting on average from one to three weeks.
  The data will be recorded as continuous variables (number of days). It will be summarized using descriptive statistics (mean ± standard deviation or median and interquartile range). It is used as one of indicators of the severity of the disease, and the data will be compared between groups of participants with different types of complicated community-acquired pneumonia, different vaccinal status and also different causative agents.
  Its relation to complications, surgical treatment, fatal outcome and incomplete radiological resolution on follow-ups will be analyzed.
Number of participants in whom intrapleural fibrinolytics were administered | from hospital admission to discharge, lasting on average from one to three weeks.
  The data will be recorded as categorical variables (two categories, with and without intrapleural fibrinolytics).
  It will be expressed as percentage of all participants. The data will be compared between groups of participants with different types of complicated community-acquired pneumonia, different vaccinal status and also different causative agents.
  Its relation to complications, surgical treatment, hospitalization length, fatal outcome and incomplete radiological resolution on follow-ups will be analyzed.
Number of participants in whom surgical treatment was performed | from hospital admission to discharge, lasting on average from one to three weeks.
  The data will be recorded as categorical variables (three categories defining different types of surgical approach).
  It will be expressed as percentage of all participants. The data will be compared between groups of participants with different types of complicated community-acquired pneumonia, different vaccinal status and different causative agents. Statistical analysis to test correlation between surgical treatment and complications, hospitalization length, fatal outcome and incomplete radiological resolution on follow-ups will be performed.
Number of patients with complications | from hospital admission to discharge, lasting on average from one to three weeks.
  The data will be recorded as categorical variables (different categories for each complication).
  It will be expressed as percentages of all participants, and is used as one of indicators of severity of the disease. The data will be compared between groups of participants with different types of complicated community-acquired pneumonia, different vaccinal status and also different causative agents. Difference in complication frequency will be compared between participants who were and were not treated with systemic corticosteroids, as well as participants in whom surgical treatment was and was not done.
  Its relation to hospitalization length, fatal outcome and incomplete radiological resolution on follow-ups will be analyzed.
Number of patients with fatal outcome of the disease | from hospital admission to discharge, lasting on average from one to three weeks.
  The data will be collected as categorical variables (categories for fatal and non-fatal outcome).
  It will be expressed as percentage of total number of participants, and is used as one of indicators of severity of the disease. The data will be compared between groups of participants with different types of complicated community-acquired pneumonia, different vaccinal status and also different causative agents.
Radiological resolution on follow-ups | Follow-ups at 3, 6 and 12 months after discharge if available.
  The data will be recorded as categorical variables (two categories regarding to complete radiological resolution and no complete resolution).
  It will be expressed as percentage of all participants. The data will be compared between groups of participants with different types of complicated community-acquired pneumonia, vaccinal status and also different causative agents, surgical treatment and intrapleural fibrinolytics.

CONTACTS AND LOCATIONS:
Locations (1):
- IMotherChildHealth, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No